CLINICAL TRIAL: NCT01348061
Title: Experimental Medicine Study to Evaluate the Kinetics of Cerebrospinal Fluid Biomarkers in Subjects With Alzheimer's Disease and Progressive Supranuclear Palsy Compared to Healthy Subjects Using a Heavy Water Labeling Method
Brief Title: Evaluating Cerebrospinal Fluid Biomarkers in Alzheimer's, Progressive Supranuclear Palsy Subjects, and Controls
Status: Completed | Type: Observational
Sponsor: KineMed (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Salena Killion, Director of Clinical Studies, KineMed
Other Study IDs: CN167001
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer Disease; Progressive Supranuclear Palsy
Keywords: Alzheimers Disease; Progressive Supranuclear Palsy; CSF; Cerebrospinal Fluid; Biomarker; Heavy Water; Cargo proteins
MeSH Terms: conditions — Alzheimer Disease; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Elderly Healthy Control (EHV): No clinically significant deviation from healthy in medical history, physical examination, ECGs, MRI and clinical laboratory determinations for their respective age group.
- Progressive Supranuclear Palsy (PSP): A diagnosis of possible or probable PSP according to clinical criteria of National Institute of Neurologic Diseases and Stroke - the Society for PSP plus a MRI at screening to exclude other potential causes of parkinsonism as well as a mild-to-moderate stage of disease severity according to a score of 1 to 3 in Golbe Staging System.
- Alzheimer's Disease (AD): A diagnosis of probable AD Based on the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association and The Diagnostic and Statistical Manual of Mental Disorders as determined by a mini-mental state examination (MMSE) score of 16 to 26, inclusive.

SUMMARY:
This is an experimental medicine study to evaluate the kinetics of cerebrospinal fluid (CSF) biomarkers in subjects with Alzheimer's disease (AD) or progressive supranuclear palsy (PSP) compared to healthy controls using a heavy water (2H2O) labeling method. This study is exploring the time profile of appearance and disappearance of pulse deuterium-labeled cargo proteins in CSF of subjects with AD and/or PSP, which is different from healthy controls, due to deficits in fast axonal transport.

DETAILED DESCRIPTION:
Primary Objective:

To compare the time profile of appearance and disappearance in CSF of pulse deuterium-labeled chromogranin B, sAPPα and β-Trace in AD and PSP subjects compared to healthy controls.

Secondary Objectives:

* To measure body water enrichment of deuterium in saliva and plasma (2H-enrichment (%))
* To explore the effect of age on the kinetics of deuterium labeling of CSF biomarkers
* To assess intra and inter subject variability of deuterium-labeling of chromogranin B, sAPPα and β-Trace

Subjects will undergo screening evaluations to determine eligibility prior to heavy water (2H20) administration. Eligible subjects will be admitted to the clinical facility on Day -1. On Day 1, subjects will ingest small doses of 2H20 during their inpatient stay. They will also drink 2H20 for 7 more days. Subjects will undergo two lumbar punctures (LPs) for CSF samples. Subjects will return to the study site approximately 7 days after the last LP (or early termination) for a follow-up assessment and discharge.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Body Mass Index of 18-32.
* Subjects can have common non-neurological age-related disorders (hypertension, diabetes) and on stable medication for the last 3 months.
* Screening score of < 4 on the Modified Hachinski Ischemia Scale.
* Women not of childbearing potential and men.
* Women with negative pregnancy test prior to starting heavy water and not breastfeeding.

AD

* Diagnosis of probable AD.
* Mild to moderate disease severity according to mini-mental state examination score (MMSE) of 16-26.
* Documented cognitive decline began 6 months prior to screening.
* On stable doses of approved AD medications for 2 months prior to screening.
* Non-medicated AD subjects are free of AD medications for 2 months prior to screening.
* Mild to moderate white matter disease and up to 2 lacunar infarcts acceptable as determined by brain MRI at screening.
* Investigator determines subjects to be medically stable and physically able to complete the study.
* Minimum of 6 years of education and able to read, write and communicate effectively.
* Adequate hearing, vision, and language skills.
* Subjects and their caregivers must agree to the dosage regimens and procedures, report for scheduled visits, and communicate with study personnel.

PSP

* Diagnosis of probable PSP.
* Brain MRI at screening excluding potential causes of parkinsonism, especially cerebrovascular and space occupying lesions.
* Mild-to-moderate stage of disease severity by a Golbe Staging System score of 1-3.
* Subjects and their caregivers must agree to the dosage regimens and procedures, report for scheduled visits, and communicate with study personnel.
* Currently on stable doses of PSP medications for 2 months prior to screening.
* Investigator determines subjects to be medically stable and able to complete the study.
* Minimum of 6 years of education and able to read, write and communicate effectively.
* Adequate hearing, vision, and language skills.

EHV

* No clinically significant deviation from healthy for their age group.
* No subjective or objective memory loss.
* MMSE score of 28 to 30.

Exclusion Criteria:

* Diseased subjects with a medical condition (not AD or PSP) that could contribute to the subjects dementia or Parkinsonism.
* History of pallidotomy, thalamotomy, active DBS or fetal tissue transplant.
* Any significant acute or chronic illness.
* Major surgery within 4 weeks of Day 1.
* Blood/plasma donation to a blood bank or a clinical study (except a screening visit) within 4 weeks of Day 1.
* Blood transfusion within 4 weeks of Day 1.
* Inability to be venipunctured.
* Inability to be lumbar punctured or contraindications to lumbar puncture or epidurals.
* > 10 cigarettes/day.
* Recent drug or alcohol abuse or positive urine screen for drugs of abuse.
* Subjects deemed inappropriate to undergo a MRI.
* Any medical, psychiatric or social reason as determined by the investigator.
* AD subjects with a history of CSF or amyloid imaging studies not consistent with Alzheimer's pathology.
* Healthy subjects with a history of CSF or amyloid imaging studies consistent with Alzheimer's pathology.
* Allergies to local anesthetics.
* Any significant drug allergy.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AD, PSP and EHV subjects will be recruited via Contract Research Organizations (CROs). Recruitment efforts will target the general population residing in communities in proximity to the CROs.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Biomarker Measures | Up to 32 days
  o Levels of deuterium-labeled chromogranin B, sAPPα and β-Trace in CSF

SECONDARY OUTCOMES:
Biomarker Measures | Up to 32 days
  o Body water enrichment of deuterium in saliva and plasma (2H-enrichment(%))

CONTACTS AND LOCATIONS:
Overall Officials: Marc K Hellerstein, M.D., Ph.D., Study Director — KineMed
Locations (3):
- United States (3):
  - Parexel, Glendale, California
  - Memory Enhancement Centers of America Inc., Eatontown, New Jersey
  - Worldwide Clinical Trials, San Antonio, Texas

REFERENCES:
- See also: Related Info — http://www.kinemed.com